CLINICAL TRIAL: NCT01160237
Title: Immunogenicity and Safety of Fluarix™/ Influsplit SSW® 2010/2011 or Pandemrix™
Brief Title: Study to Evaluate the Immune Response and the Safety of Fluarix TM/ Influsplit SSW® 2010/2011 or Pandemrix TM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated for logistic reasons not related to safety or efficacy of the vaccine.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114454
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-09

CONDITIONS: Influenza
Keywords: H1N1; Pandemrix; Fluarix; Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (3):
- Group A (Experimental): Subjects previously vaccinated with a vaccine against the pandemic H1N1 strain
  Interventions: Biological: PandemrixTM
- Group B (Experimental): Subjects previously vaccinated with a vaccine against the pandemic H1N1 strain
  Interventions: Biological: FluarixTM/ Influsplit SSW® 2010/2011
- Group C (Active Comparator): Subjects not previously vaccinated with a vaccine against the pandemic H1N1 strain
  Interventions: Biological: FluarixTM/ Influsplit SSW® 2010/2011

INTERVENTIONS:
Biological: PandemrixTM — One dose intramuscular injection
  Arms: Group A
Biological: FluarixTM/ Influsplit SSW® 2010/2011 — One dose intramuscular injection
  Arms: Group B; Group C

SUMMARY:
The aim of this study is to evaluate the immune response and the safety of one injection of FluarixTM/ Influsplit SSW® 2010/2011 or Pandemrix TM in subjects who had received a single Pandemrix TM dose at least 6 months preceding study inclusion. Subjects never vaccinated with any H1N1 pandemic vaccine will be enrolled as control.

This Protocol Posting has been updated following Amendment of the Protocol, July 2010. The impacted section is entry criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol. Specific attention should be given to the compliance potential of subjects with suspected or known drug and alcohol abuse.
* Subjects who have received one dose of Pandemrix at least 6 month before enrolment, to be enrolled in the Groups A or B OR subjects who have not been previously vaccinated with a vaccine against the pandemic H1N1 strain at all, to be enrolled in group C.
* A male or female 18 years and above at the time of enrolment.
* Written informed consent obtained from the subject.
* Healthy subjects or free of acute aggravation of the health status as established by physical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Administration of any influenza vaccine within 6 month prior to vaccination in this study.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature ≥ 37.5ºC, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer, within the past 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Chronic administration of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period..
* Any administration of a long-acting immune-modifying drug (within 3 months before study start, or a planned administration during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Administration of any vaccines within 30 days before vaccination.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions from study inclusion up to 2 months after completion of the vaccination series.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (5):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Pandemrix Group: Subjects previously vaccinated with Pandemrix received 1 dose of Pandemrix.
- Fluarix Group: Subjects previously vaccinated with Pandemrix received one dose of Fluarix.
- Control Group: Subjects not previously vaccinated with Pandemrix received one dose of Fluarix.
Period: Overall Study
Arm/Group | Pandemrix Group | Fluarix Group | Control Group
Started | 4 | 3 | 0
Completed | 4 | 3 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pandemrix Group | Fluarix Group | Control Group | Total
Number analyzed (Participants) | 4 | 3 | 0 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.50) | 55.3 (18.80) |  | 58.7 (13.16)
Gender [Number; unit: subjects]
  Female | 3 | 2 |  | 5
  Male | 1 | 1 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies for Each Vaccine Strain, in Subjects Aged 18-60 and Above 60 Years
Time Frame: 21 days after vaccination
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | Pandemrix Group | Fluarix Group | Control Group
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Solicited Local and General Symptoms
Time Frame: During 7 days (Day 0 - Day 6) after vaccination
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | Pandemrix Group | Fluarix Group | Control Group
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Time Frame: During 31 days (Day 0 - Day 30) after vaccination
Population: The analysis was performed on the total vaccinated cohort. No subjects were enrolled in the Control Group by the time the study was prematurely terminated.
Measure: Number; unit: subjects
Arm/Group | Pandemrix Group | Fluarix Group | Control Group
Number analyzed (Participants) | 4 | 3 | 0
subjects | 0 | 2 |

4. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events
Time Frame: During the whole study period (Day 0 - Day 182)
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Pandemrix Group | Fluarix Group | Control Group
Number analyzed (Participants) | 4 | 3 | 0
subjects | 1 | 0 |

5. Secondary Outcome: Potential Immune Mediated Diseases
Time Frame: During the whole study period (Day 0 - Day 182)
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | Pandemrix Group | Fluarix Group | Control Group
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Humoral Immune Response in Terms of HI Antibodies Against Each Vaccine Strain, at Different Timepoints in Subjects Aged 18-60 and Above 60 Years
Time Frame: At Days 0, 7 and 182
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | Pandemrix Group | Fluarix Group | Control Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pandemrix Group | Fluarix Group | Control Group
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 2/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pandemrix Group (N=4) | Fluarix Group (N=3) | Control Group (N=0)
femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pandemrix Group (N=4) | Fluarix Group (N=3) | Control Group (N=0)
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Only 7 subjects were enrolled in either the Pandemrix Group or the Fluarix Group and none in the Control Group since the study was terminated prematurely. Therefore most outcome measures (except unsolicited AEs and SAEs) were not analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.